CLINICAL TRIAL: NCT01807442
Title: Developing a Positive Psychology Intervention to Improve Cardiac Health Behaviors: Qualitative Research Phase
Brief Title: Positive Psychology to Improve Cardiac Health Behaviors
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director of Inpatient Psychiatric Unit, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011P002729; 1R01HL113272-01A1 (NIH)
Record Dates: First submitted 2013-03-04; First posted 2013-03-08 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Acute Coronary Syndrome; Emotions; Patient Compliance
Keywords: Acute Coronary Syndrome; Positive Psychology; Adherence to Health Behaviors
MeSH Terms: conditions — Acute Coronary Syndrome; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimal adherence (Other): Participants receive the qualitative interview and adherence intervention.
  This arm includes participants with scores of greater than or equal to 15 on the Medical Outcomes Study Specific Adherence Scale. This scale ranges from a score of 3 (extremely low adherence to health behaviors) to a score of 18 (extremely high adherence to health behaviors). A score of greater than or equal to 15 suggests optimal adherence to health behaviors.
  Interventions: Other: Qualitative Interview and Adherence
- Sub-optimal adherence (Other): Participants receive the qualitative interview and adherence intervention.
  This arm includes participants with scores of less than 15 on the Medical Outcomes Study Specific Adherence Scale. This scale ranges from a score of 3 (extremely low adherence to health behaviors) to a score of 18 (extremely high adherence to health behaviors). A score of less than 15 suggests sub-optimal adherence to health behaviors.
  Interventions: Other: Qualitative Interview and Adherence

INTERVENTIONS:
Other: Qualitative Interview and Adherence — All participants receive the same intervention. The intervention involves two qualitative interviews per participant. The first interview occurs in the hospital, and the second interview occurs at 12 weeks. Participants also receive a pill bottle that tracks when they take their aspirin. They will also receive a step counter to use for two weeks at the end of the study.

SUMMARY:
The purpose of the study is to understand peoples' positive emotions, like how optimistic or grateful they feel, after they have had a heart problem. The investigators want to determine whether positive emotions affect peoples' ability to follow recommendations, like following a healthy diet, exercising, and taking medication.

DETAILED DESCRIPTION:
The investigators aim to develop a novel positive psychology intervention that is adapted for patients hospitalized for an acute coronary syndrome (ACS). A treatment cultivating positive emotions in this vulnerable population could provide broad and significant health benefits, and may have distinct-and more powerful-effects than simply attempting to dampen negative emotions.

In this study, the investigators will use mixed methods (qualitative and quantitative) to take the first step towards developing such a treatment, with a major focus on the qualitative aspects of the patient assessments/interviews.

In this project, the investigators hope to do the following:

1. Identify, through qualitative research, deficits in positive emotional and cognitive states prior to, during, and after cardiac admission: What positive emotions are lacking in hospitalized ACS patients?
2. Explore strategies to enhance positive emotional and cognitive states in ACS patients.
3. Identify links between these positive states and health behavior (diet, physical activity, and medication).
4. Identify other barriers to compliance with health behaviors. What other factors adversely influence compliance with health behaviors in this population?
5. Use quantitative measures of positive affect to ensure that the investigators are adequately capturing information about optimism and other positive states
6. Develop a preliminary positive psychology-based intervention using the above information
7. Explore the feasibility of using methods to objectively measure aspirin adherence and physical activity in this population.

To accomplish these goals, the investigators will interview 30 ACS patients during admission to the inpatient cardiac unit and 12 weeks after discharge. The investigators will identify 15 patients who demonstrate suboptimal adherence as reported by the Medical Outcomes Study Specific Adherence Scale (MOS-SAS) and 15 patients who demonstrate good adherence to health-related behaviors.

For these interviews, the investigators will first ask about positive emotional states that patients have experienced. the investigators will then inquire about potential ideas for increasing these positive emotional states by asking patients what has worked for them in the past and what they have noticed seems to work for others. The investigators will also describe some positive psychology exercises to the patients and ask whether they think those exercises would be effective at increasing positive emotional states. Next, the investigators will ask about health behaviors in which the patient has engaged. The investigators will explore the relationship between these behaviors and positive emotional states. Finally, the investigators will explore with patients some barriers to completing health behaviors and solicit suggestions for overcoming or mitigating these barriers.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Massachusetts General Hospital cardiac floors (Ellison 9, 10, 11)
* Age 18 or older
* Admitted with myocardial infarction or unstable angina
* Score of less than 15 --OR-- greater than or equal to 15 on the adherence scale
* Ability to read and write in English

Exclusion Criteria:

* Cognitive deficits as assessed by a 6-item screen
* Medical conditions that prevent interviewing or are likely to lead to death within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Deficits in positive affect | 12 weeks
  Qualitative data:
  The investigators will extract information from 2 quantitative interviews to learn about participants' deficits in positive affect.
  Quantitative data:
  Life Orientation Test-Revised, Positive And Negative Affect Scale, Hospital Anxiety and Depression Scale.
Barriers to health behaviors | 12 weeks
  Qualitative data:
  The investigators will extract information from 2 qualitative interviews to learn about participants' barriers to completing health behaviors.
  Quantitative data:
  Participants will receive a pill bottle that tracks when they take their aspirin. Participants will also receive a step counter to wear for two weeks.

SECONDARY OUTCOMES:
Changes in positive affect | Change from baseline positive affect at 12 weeks
  Qualitative data:
  The investigators will compare information from the 2 qualitative interviews to learn about participants' changes in positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States